CLINICAL TRIAL: NCT04380025
Title: The Effects of Mirtogenol® With Bimatoprost on Intraocular Pressure in Hispanics With Open-Angle Glaucoma: A Double-Blind, Randomized Controlled Trial
Brief Title: Mirtogenol and Bimatoprost on IOP in Hispanics With Open-Angle Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Jorge R. Miranda-Massari, Professor, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A4570119
Record Dates: First submitted 2020-02-27; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-03

CONDITIONS: Glaucoma
Keywords: bimatoprost; hispanic; Mirtogenol; bilberry; Pycnogenol
MeSH Terms: conditions — Glaucoma | interventions — Vaccinium myrtillus extract; pycnogenols; Lactose

STUDY DESIGN:
Intervention Model Description: A prospective, parallel-group, double-blind, randomized placebo-controlled clinical trial will be conducted with an estimated 72 primary open-angle glaucoma patients. A double blind RCT was chosen to minimize bias and yield similar groups with the same prognostic at baseline to avoid compromising the validity of the study results. The primary efficacy endpoint of the study will be IOP and the secondary endpoint will be the safety analysis.
Who Masked: Participant, Care Provider
Masking Description: This is a double blind study. The participant and the medical care provider will not know the identity of the placebo or study product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirtogenol (Experimental): In addition of conventional treatment with glaucoma ophtalmic drop medication (bimatoprost) the experimental group will also take Mirtogenol. Mirtogenol is a dietary supplement composed of bilberry and pycnogenol which are botanical compounds with antioxidant properties. The active components of bilberry are flavonoid anthocyanosides (anthocyanins). Anthocyanosides are the only flavonoids able to reach the eye as a target organ in experimental animals. Unchanged anthocyanosides demonstrated after oral administration that it is absorbed and distributed into ocular tissues, showing its ability to pass through the blood-aqueous and blood retinal barriers.6
  Interventions: Dietary Supplement: Experimental: Oral Mirtogenol
- Lactose based Placebo (Placebo Comparator): In addition of conventional treatment with glaucoma ophtalmic drop medication (bimatoprost) this control group will also take an identical placebo. This placebo is a inactive lactose based product of the same color and size capsule.
  Interventions: Dietary Supplement: Placebo of oral Dietary supplement

INTERVENTIONS:
Dietary Supplement: Experimental: Oral Mirtogenol — The experimental arm is Oral Mirtogenol dietary supplement, one capsule daily in addition to bimatoprost ophthalmic drops with primary open angle glaucoma
  Other Names: Bilberry with pycnogenol
  Arms: Mirtogenol
Dietary Supplement: Placebo of oral Dietary supplement — This is the oral placebo of the supplement (control) un daily capsule in addition to the bimatoprost ophtalmic drops
  Other Names: lactose and food grade dyes
  Arms: Lactose based Placebo

SUMMARY:
A prospective, parallel-group, double-blind, randomized placebo-controlled clinical study will be conducted with an estimated 72 participants. The objective of this study is to determine if Mirtogenol has an additive effect on the reduction of intraocular pressure when combined with bimatoprost in the Hispanic population with primary open angle glaucoma. Baseline clinical data will be collected for each participant and they will be randomized 1:1 to a treatment group (bimatoprost 0.01% and Mirtogenol) or control group (bimatoprost 0.01% and placebo). Efficacy and safety of Mirtogenol will be measured during the 24 week study. Participants will be evaluated in five visits: screening and baseline, week 4, week 8, week 12 and week 24. The tests that will be performed include visual acuity, visual field evaluation, applanation tonometry, optical coherence tomography (OCT), and pachymetry. Side effects or adverse effects will be reported and evaluated by the ophthalmologist at each visit to access the safety of Mirtogenol. The primary efficacy endpoint of intraocular pressure (IOP) will be compared using a t-test and will have an 80% probability to detect a difference between treatments at a 0.05 significance level.

DETAILED DESCRIPTION:
METHODOLOGY AND STUDY DESIGN A prospective, parallel-group, double-blind, randomized placebo-controlled clinical trial will be conducted with an estimated 72 primary open-angle glaucoma patients. A double blind RCT was chosen to minimize bias and yield similar groups with the same prognostic at baseline to avoid compromising the validity of the study results. The primary efficacy endpoint of the study will be IOP and the secondary endpoint will be the safety analysis. Qualifying participants will be evaluated for inclusion and exclusion criteria by their ophthalmologist (Dr. Marino Blasini) and informed about the study objectives. If they agree to participate, relevant baseline clinical data will be collected for each participant and they will be assigned to a treatment or a control group by stratified randomization based on their age, intraocular pressure and cup-to-disk ratio. This stratified randomization will allow comparability of randomized study groups at baseline. Participants will be randomized in a 1:1 ratio to treatment group (bimatoprost 0.01% and Mirtogenol®) or control group (bimatoprost 0.01% and placebo) and be assigned a participant ID number. Once the randomization process has concluded, participants will be notified to pass by the office to receive the product and to start using the Mirtogenol® or placebo the next day. Both Mirtogenol® and placebo bottles will label drug of study and be registered with a number identification for each patient. Mirtogenol and the placebo will be stored in a destinated area in the primary investigator's pharmacy under a cool, dry environment that protects them from extreme temperature changes and light. Oral and written instructions on drug regimen, including route of administration, frequency, proper storage and mode of administer will be provided. The groups will self-instill one drop of bimatoprost 0.01% in the affected eye(s) once daily as instructed by the ophthalmologist. In addition, participants will use one (1) capsule of Mirtogenol® or one (1) placebo capsule orally daily in the morning with food. Mirtogenol® will be funded by Life Extension Clinical Research, Inc. Placebo capsules will be similar in appearance, size, and route of administration to Mirtogenol®. The study will have five visits: screening and baseline, week 4, week 8, week 12 and week 24 of approximate 30-60 minutes of duration and an addition visit for pickup of the product after the randomization process. An ophthalmological evaluation will be conducted by a glaucoma specialist at each visit. At the baseline visit, the following tests will be performed: visual acuity, visual field evaluation, applanation tonometry, optical coherence tomography (OCT), and pachymetry. At week 4, and week 8 the following tests will be performed: visual acuity and applanation tonometry. At week 12, the following tests will be performed: visual acuity, visual field evaluation and applanation tonometry. At week 24, assessments will include the following: visual acuity, visual field evaluation, applanation tonometry, optical coherence tomography and pachymetry. The same equipment will be used throughout the study for measurement consistency. Each test will be measured in the morning and the patient will be resting, sitting for at least 10 minutes before measurement. The tests will always be performed by the same person to rule out variations. At each visit, the IOP will be measured twice, with 10-minute intermissions between measurements, and mean values will be recorded. If only one eye is determined eligible as trial eye (meeting the diagnostic criteria for glaucoma), then all assessments will be performed only for the trial eye. If both eyes are eligible, only the eye with highest baseline mean IOP will be included in the statistical analysis. Patients will be instructed not to take any medications within two hours before measurements. Any therapy considered necessary for the patient's welfare will be given at the discretion of the treating physician and will be documented. Safety measures include non-invasive techniques, standard of care treatment during the duration of the study, ophthalmological evaluations and assessment tests. Side effects or adverse effects will be reported and evaluated by the ophthalmologist at each visit and if deemed necessary the trial medication (Mirtogenol® or matching placebo) will be discontinued and therapy adjusted as appropriate by the clinician. Adverse effects will be recorded at each study visit as well as the probability of possible association of the adverse effects to the treatment. Compliance will be reinforced with daily reminder for a month by email or text messages and then weekly reminders until the termination of the study. A monthly calendar will be provided to keep track of doses and possible miss doses. Patient must bring their supplement or placebo bottles and monthly track calendar to each visit and a pill count will be performed. Participants will be contacted one month after discontinuing the trial medication to assess for any prior changes or side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma (POAG)
* over 21 yrs
* Self identified as hispanic
* Current glaucoma treatment regimen of monotherapy with bimatoprost 0.01% applie into affected eye(s) once daily and with stable IOP less or equal to 21 mmHG

Exclusion Criteria:

* Less than 21 year old
* Pregnant women (self-reported) or those who are planning to become pregnant in the next six (6) months (There is insufficient reliable information available about the safety of Mirtogenol® when used in medicinal amounts during pregnancy and lactation)
* Women who are breastfeeding (There is insufficient reliable information available about the safety of Mirtogenol® when used in medicinal amounts during pregnancy and lactation)
* Individuals with cardiovascular diseases that have required medical intervention in the past three (3) months
* Patients that required any kind of surgery, radiotherapy or chemotherapy in the past three (3) months
* Patients with advanced glaucoma with a cup to disk ratio > 0.9, previous glaucoma surgeries or other abnormalities of the eye that affect the visual pathway

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Change in intraocular pressure (IOP) | Participants will be evaluated in five visits: screening and baseline, week 4, week 8, week 12 and week 24.
  intraocular pressure (IOP) will be compared using a t-test and will have an 80% probability to detect a difference between treatments at a 0.05 significance level.

SECONDARY OUTCOMES:
Change in the Tolerance of the experimental supplement | 24 weeks
  The safety of the combination of Mirtogenol® with bimatoprost will be evaluated, specifically, recording gastrointestinal or neurological symptoms if any.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge R Miranda, Pham.D., Principal Investigator — School of Pharmacy, University of Puerto Rico, Medical Sciences Campus
Locations (1):
- University of Puerto Rico, Medical Sciences Campus, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steigerwalt RD Jr, Belcaro G, Morazzoni P, Bombardelli E, Burki C, Schonlau F. Mirtogenol potentiates latanoprost in lowering intraocular pressure and improves ocular blood flow in asymptomatic subjects. Clin Ophthalmol. 2010 May 14;4:471-6. doi: 10.2147/opth.s9899. PMID 20505841
- [Background] Gizzi C, Torino-Rodriguez P, Belcaro G, Hu S, Hosoi M, Feragalli B. Mirtogenol(R) supplementation in association with dorzolamide-timolol or latanoprost improves the retinal microcirculation in asymptomatic patients with increased ocular pressure. Eur Rev Med Pharmacol Sci. 2017 Oct;21(20):4720-4725. PMID 29131240
- [Result] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- [Result] Distelhorst JS, Hughes GM. Open-angle glaucoma. Am Fam Physician. 2003 May 1;67(9):1937-44. PMID 12751655
- [Result] Munemasa Y, Kitaoka Y. Molecular mechanisms of retinal ganglion cell degeneration in glaucoma and future prospects for cell body and axonal protection. Front Cell Neurosci. 2013 Jan 9;6:60. doi: 10.3389/fncel.2012.00060. eCollection 2012. PMID 23316132
- [Result] Steigerwalt RD, Gianni B, Paolo M, Bombardelli E, Burki C, Schonlau F. Effects of Mirtogenol on ocular blood flow and intraocular hypertension in asymptomatic subjects. Mol Vis. 2008 Jul 10;14:1288-92. PMID 18618008

DOCUMENTS (2):
  • Study Protocol (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT04380025/Prot_000.pdf
  • Informed Consent Form (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT04380025/ICF_001.pdf